CLINICAL TRIAL: NCT04833686
Title: The Effect of Music and Environmental Noise Isolation on Bronchiolitis Severity in Hospitalized Children: a Randomized Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, noa ziv, MD, Schneider Children's Medical Center, Israel
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0755-17
Record Dates: First submitted 2021-03-29; First posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Bronchiolitis
Keywords: Double blind randomized controlled study; Prospective
MeSH Terms: conditions — Bronchiolitis | interventions — SIR1 protein, S cerevisiae

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sonata for 2 pianos in D major, K.488 by Mozart (Active Comparator): An Mp3 player, upload with music by Mozart. Music was played using headphones suitable and approved for use in children.
  Interventions: Behavioral: Mozart
- Instrumental music ("To the Point", by Dean Evenson & Tom Barabas) (Active Comparator): An Mp3 player, upload with instrumental music. Music was played using headphones suitable and approved for use in children.
  Interventions: Behavioral: Instrumental music
- Silence (Active Comparator): An Mp3 player, upload with silence. Silence was played using headphones suitable and approved for use in children.
  Interventions: Behavioral: Silence

INTERVENTIONS:
Behavioral: Mozart — Music composed by Mozart, a musical piece 24 minutes long.
  Arms: Sonata for 2 pianos in D major, K.488 by Mozart
Behavioral: Instrumental music — Instrumental music , a musical piece 24 minutes long
  Arms: Instrumental music ("To the Point", by Dean Evenson & Tom Barabas)
Behavioral: Silence — Silence, a piece 24 minutes long.
  Arms: Silence

SUMMARY:
Bronchiolitis is an infectious disease, with no effective treatment. Music and Mozart's works specifically, has been shown to have a positive effect on physiological parameters, while environmental noise is considered to be harmful. We aimed to evaluate the short-time effect of listening to music and detachment from environmental noise on the severity of bronchiolitis in hospitalized children.

DETAILED DESCRIPTION:
MP3 player devices were uploaded with 3 different pieces: 1) sonata for 2 pianos in D major, K.488 by Mozart (2) instrumental music ("To the Point", by Dean Evenson & Tom Barabas) and (3) silence. All music or silence pieces were identical in length (24 minutes in accordance to the duration of the sonata).

Music fragments were played using headphones suitable and approved for use in children - GSI (Grason-Standler) Insert Earphone TIP-50 (50 ohm) (Grason Standler Inc. Madison, WI, USA). Sound frequency and volume were adjusted to the age appropriate values33 Children were randomly divided into 3 groups according to the type of intervention. Randomization, numbering of the MP3 players and coding of the content were done by a research coordinator not involved in evaluation of the patients nor in analysis of the results.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 0-24 months, with the clinical diagnosis of bronchiolitis.

Exclusion Criteria:

* Children who failed neonatal hearing screening or in whom the results of the screening were not available were excluded from the study.
* Children who were not able to maintain listening for at least 10 minutes were excluded from data analysis

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Change in disease severity | Evaluation was done before music playing and immediately after the end of the music session (At 0 minutes time, and at a maximum time of 24 minutes from the beginning of intervention - which is the length of the musical piece).
  Evaluated by Modified Tal Score (Respiratory rate, O2 saturation, use of accessory respiratory muscles, breath sounds: wheezing)

CONTACTS AND LOCATIONS:
Overall Officials: Noa Ziv, MD, Principal Investigator — Schneider Children's Medical Center, Israel
Locations (1):
- Schneider Children's Medical Center of Israel, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Friedman JN, Rieder MJ, Walton JM; Canadian Paediatric Society, Acute Care Committee, Drug Therapy and Hazardous Substances Committee. Bronchiolitis: Recommendations for diagnosis, monitoring and management of children one to 24 months of age. Paediatr Child Health. 2014 Nov;19(9):485-98. doi: 10.1093/pch/19.9.485. PMID 25414585
- [Background] Ralston SL, Lieberthal AS, Meissner HC, Alverson BK, Baley JE, Gadomski AM, Johnson DW, Light MJ, Maraqa NF, Mendonca EA, Phelan KJ, Zorc JJ, Stanko-Lopp D, Brown MA, Nathanson I, Rosenblum E, Sayles S 3rd, Hernandez-Cancio S; American Academy of Pediatrics. Clinical practice guideline: the diagnosis, management, and prevention of bronchiolitis. Pediatrics. 2014 Nov;134(5):e1474-502. doi: 10.1542/peds.2014-2742. PMID 25349312
- [Background] Ricci V, Delgado Nunes V, Murphy MS, Cunningham S; Guideline Development Group and Technical Team. Bronchiolitis in children: summary of NICE guidance. BMJ. 2015 Jun 2;350:h2305. doi: 10.1136/bmj.h2305. No abstract available. PMID 26037525
- [Background] Kassis I, Srugo I, Srur S, Horowitz Y, Almagor T, Wolf D, Kra-Oz Z, Kennes Y, Rishpon S, Miron D. [The burden and outcomes of acute bronchiolitis among young children hospitalized in Israel]. Harefuah. 2009 Nov;148(11):748-51, 795, 794. Hebrew. PMID 20027974
- [Background] Kou M, Hwang V, Ramkellawan N. Bronchiolitis: From Practice Guideline to Clinical Practice. Emerg Med Clin North Am. 2018 May;36(2):275-286. doi: 10.1016/j.emc.2017.12.006. Epub 2018 Feb 10. PMID 29622322
- [Background] Hasegawa K, Tsugawa Y, Brown DF, Mansbach JM, Camargo CA Jr. Trends in bronchiolitis hospitalizations in the United States, 2000-2009. Pediatrics. 2013 Jul;132(1):28-36. doi: 10.1542/peds.2012-3877. Epub 2013 Jun 3. PMID 23733801
- [Background] Vaajoki A, Kankkunen P, Pietila AM, Vehvilainen-Julkunen K. Music as a nursing intervention: effects of music listening on blood pressure, heart rate, and respiratory rate in abdominal surgery patients. Nurs Health Sci. 2011 Dec;13(4):412-8. doi: 10.1111/j.1442-2018.2011.00633.x. Epub 2011 Sep 8. PMID 21902776
- [Background] Golino AJ, Leone R, Gollenberg A, Christopher C, Stanger D, Davis TM, Meadows A, Zhang Z, Friesen MA. Impact of an Active Music Therapy Intervention on Intensive Care Patients. Am J Crit Care. 2019 Jan;28(1):48-55. doi: 10.4037/ajcc2019792. PMID 30600227
- [Background] Pauwels EK, Volterrani D, Mariani G, Kostkiewics M. Mozart, music and medicine. Med Princ Pract. 2014;23(5):403-12. doi: 10.1159/000364873. Epub 2014 Jul 19. PMID 25060169
- [Background] Warren JD. Variations on the musical brain. J R Soc Med. 1999 Nov;92(11):571-5. doi: 10.1177/014107689909201108. No abstract available. PMID 10703494
- [Background] Loomba RS, Arora R, Shah PH, Chandrasekar S, Molnar J. Effects of music on systolic blood pressure, diastolic blood pressure, and heart rate: a meta-analysis. Indian Heart J. 2012 May-Jun;64(3):309-13. doi: 10.1016/S0019-4832(12)60094-7. PMID 22664817
- [Background] Uchiyama M, Jin X, Zhang Q, Hirai T, Amano A, Bashuda H, Niimi M. Auditory stimulation of opera music induced prolongation of murine cardiac allograft survival and maintained generation of regulatory CD4+CD25+ cells. J Cardiothorac Surg. 2012 Mar 23;7:26. doi: 10.1186/1749-8090-7-26. PMID 22445281
- [Background] Lee JH. The Effects of Music on Pain: A Meta-Analysis. J Music Ther. 2016 Winter;53(4):430-477. doi: 10.1093/jmt/thw012. Epub 2016 Oct 19. PMID 27760797
- [Background] Tolunay T, Bicici V, Tolunay H, Akkurt MO, Arslan AK, Aydogdu A, Bingol I. Rhythm and orthopedics: The effect of music therapy in cast room procedures, a prospective clinical trial. Injury. 2018 Mar;49(3):593-598. doi: 10.1016/j.injury.2018.02.008. Epub 2018 Feb 7. PMID 29454656
- [Background] McConnell T, Porter S. Music therapy for palliative care: A realist review. Palliat Support Care. 2017 Aug;15(4):454-464. doi: 10.1017/S1478951516000663. Epub 2016 Oct 24. PMID 27772537
- [Background] Stegemann T, Geretsegger M, Phan Quoc E, Riedl H, Smetana M. Music Therapy and Other Music-Based Interventions in Pediatric Health Care: An Overview. Medicines (Basel). 2019 Feb 14;6(1):25. doi: 10.3390/medicines6010025. PMID 30769834
- [Background] Rauscher FH, Shaw GL, Ky KN. Music and spatial task performance. Nature. 1993 Oct 14;365(6447):611. doi: 10.1038/365611a0. No abstract available. PMID 8413624
- [Background] Lubetzky R, Mimouni FB, Dollberg S, Reifen R, Ashbel G, Mandel D. Effect of music by Mozart on energy expenditure in growing preterm infants. Pediatrics. 2010 Jan;125(1):e24-8. doi: 10.1542/peds.2009-0990. Epub 2009 Dec 7. PMID 19969615
- [Background] Coppola G, Toro A, Operto FF, Ferrarioli G, Pisano S, Viggiano A, Verrotti A. Mozart's music in children with drug-refractory epileptic encephalopathies. Epilepsy Behav. 2015 Sep;50:18-22. doi: 10.1016/j.yebeh.2015.05.038. Epub 2015 Jun 18. PMID 26093514
- [Background] Jenkins JS. The Mozart effect. J R Soc Med. 2001 Apr;94(4):170-2. doi: 10.1177/014107680109400404. No abstract available. PMID 11317617
- [Background] Goines L, Hagler L. Noise pollution: a modem plague. South Med J. 2007 Mar;100(3):287-94. doi: 10.1097/smj.0b013e3180318be5. PMID 17396733
- [Background] Hsu, T., Ryherd, E. E., Waye, K. P., & Ackerman, J. (2012). Noise pollution in hospitals: Impact on patients. Journal of Clinical Outcomes Management, 19(7), 301-309.
- [Background] Gupta A, Gupta A, Jain K, Gupta S. Noise Pollution and Impact on Children Health. Indian J Pediatr. 2018 Apr;85(4):300-306. doi: 10.1007/s12098-017-2579-7. Epub 2018 Jan 9. PMID 29313308
- [Background] Xyrichis A, Wynne J, Mackrill J, Rafferty AM, Carlyle A. Noise pollution in hospitals. BMJ. 2018 Nov 18;363:k4808. doi: 10.1136/bmj.k4808. No abstract available. PMID 30449734
- [Background] Stansfeld S, Clark C. Health Effects of Noise Exposure in Children. Curr Environ Health Rep. 2015 Jun;2(2):171-8. doi: 10.1007/s40572-015-0044-1. PMID 26231366
- [Background] Kramer B, Joshi P, Heard C. Noise pollution levels in the pediatric intensive care unit. J Crit Care. 2016 Dec;36:111-115. doi: 10.1016/j.jcrc.2016.06.029. Epub 2016 Jul 9. PMID 27546758
- [Background] Ryan KM, Gagnon M, Hanna T, Mello B, Fofana M, Ciottone G, Molloy M. Noise Pollution: Do We Need a Solution? An Analysis of Noise in a Cardiac Care Unit. Prehosp Disaster Med. 2016 Aug;31(4):432-5. doi: 10.1017/S1049023X16000388. Epub 2016 May 23. PMID 27211892
- [Background] Linares C, Diaz J, Tobias A, De Miguel JM, Otero A. Impact of urban air pollutants and noise levels over daily hospital admissions in children in Madrid: a time series analysis. Int Arch Occup Environ Health. 2006 Feb;79(2):143-52. doi: 10.1007/s00420-005-0032-0. Epub 2005 Sep 27. PMID 16187125
- [Background] Eze IC, Foraster M, Schaffner E, Vienneau D, Heritier H, Pieren R, Thiesse L, Rudzik F, Rothe T, Pons M, Bettschart R, Schindler C, Cajochen C, Wunderli JM, Brink M, Roosli M, Probst-Hensch N. Transportation noise exposure, noise annoyance and respiratory health in adults: A repeated-measures study. Environ Int. 2018 Dec;121(Pt 1):741-750. doi: 10.1016/j.envint.2018.10.006. Epub 2018 Oct 12. PMID 30321849
- [Background] Brown G. NICU noise and the preterm infant. Neonatal Netw. 2009 May-Jun;28(3):165-73. doi: 10.1891/0730-0832.28.3.165. PMID 19451078
- [Background] Wachman EM, Lahav A. The effects of noise on preterm infants in the NICU. Arch Dis Child Fetal Neonatal Ed. 2011 Jul;96(4):F305-9. doi: 10.1136/adc.2009.182014. Epub 2010 Jun 14. PMID 20547580
- [Background] McCallum GB, Morris PS, Wilson CC, Versteegh LA, Ward LM, Chatfield MD, Chang AB. Severity scoring systems: are they internally valid, reliable and predictive of oxygen use in children with acute bronchiolitis? Pediatr Pulmonol. 2013 Aug;48(8):797-803. doi: 10.1002/ppul.22627. Epub 2012 Sep 4. PMID 22949369
- [Background] W. J. Dixon. BMDP Statistical Software. 1993.
- [Background] Finn S, Fancourt D. The biological impact of listening to music in clinical and nonclinical settings: A systematic review. Prog Brain Res. 2018;237:173-200. doi: 10.1016/bs.pbr.2018.03.007. Epub 2018 May 1. PMID 29779734
- [Background] Guski R, Schreckenberg D, Schuemer R. WHO Environmental Noise Guidelines for the European Region: A Systematic Review on Environmental Noise and Annoyance. Int J Environ Res Public Health. 2017 Dec 8;14(12):1539. doi: 10.3390/ijerph14121539. PMID 29292769
- See also: WHO work on noise — https://www.euro.who.int/en/health-topics/environment-and-health/noise